CLINICAL TRIAL: NCT01829763
Title: Central Effects of Botulinum Toxin: Neurophysiological Study in Stroke Patients With Spastic Lower Limb
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-000600-42; 2013-02 (Other: AP HM)
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Hemiplegic Patients Post-AVC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- botox (Experimental)
  Interventions: Drug: injection botox

INTERVENTIONS:
Drug: injection botox

SUMMARY:
Spasticity is a motor disorder characterized by a velocity-dependent increase in tonic stretch reflex with exaggerated tendon jerk (Lance 1980). Patients with brain lesion often display spasticity due to the interruption of the descending pathways that control the spinal reflex networks, which results in hyperexcitability of the monosynaptic reflex triggered by stretch of the muscle spindles. Spasticity in lower limb muscle impairs the gait, especially in strokes that are the main cause of neurological disability. While 80% of the stroke survivors recover the ability to walk, the poor quality of their gait constitutes a serious handicap in daily life (Bensoussan et al. 2004; Bensoussan et al. 2006).

Local injection of Botulinum toxin (BTx) has become a mainstay of the treatment of focal spasticity, particularly in post-stroke patients. BTx weakens the excessive muscle contraction by blocking the release of acethylcholine from motoneuron terminals at the neuromuscular junction and transiently paralyzing the muscle for several months. Besides this peripheral action, BTx is assumed to have also a central effect (Curra et al. 2004; Gracies 2004; Krishnan 2005; Palomar and Mir 2012). In particular, by affecting also the fusimotor synapses on intrafusal muscles fibers (Rosales and Dressler 2010; Trompetto et al. 2008; Trompetto et al. 2006), BTx may reduce the discharge from muscle spindles, which may be indirectly responsible for functional changes in central motor mechanisms at both spinal and supraspinal levels. Animal experiments also suggested that BTx is carried by retrograde axonal transport to motoneuron soma and possibly transynaptically, and can affect the spinal cholinergic synaptic transmission in the spinal cord. Until now, electrophysiological findings are limited and controversial, probably due to the various motor disorders investigated, the physiological mechanisms tested and the different toxin injection protocols used in the few studies available (Frascarelli et al. 2011; Girlanda et al. 1997; Modugno et al. 1998; Naumann and Reiners 1997; Pauri et al. 2000; Priori et al. 1995; Wohlfarth et al. 2001). Hence, the central action of the toxin in spasticity remains uncertain.

ELIGIBILITY:
Inclusion Criteria:

* More than 18-years-old Patient
* Patient presenting a hemiplegia séquellaire of an AVC above - tentoriel dating more than 12 months
* Patient presenting a spasticité of the muscles of the leg
* Patient for him(it) ( a ) which an indication of treatment(processing) by botulinal toxin is carried(worn)
* Patient not having received from treatment(processing) by botulinal toxin at the level of the lower limb for six months
* Patient not having benefited from alcoholization or surgical gesture(movement) at the level of the lower limb for twelve months
* Spasticité focused the muscles of leg: soleus, gastrocnémiens, with score of Ashworth > or = 2 on the concerned muscles and/or the presence of a clonus on the soleus or gastrocnémiens,

Exclusion Criteria:

* Patient for him(it) ( a ) which the upright posture and/or the walking(step) are impossible
* Patient presenting a contraindication to the use of the botulinal toxin
* Patient presenting a contraindication to the use of the intramuscular way
* Patient susceptible not to participate in the totality of the study
* Woman pregnant or susceptible to be pregnant during the year
* Patient who can not give himself(itself) his consent (held(detained), major under guardianship)
* Patient incapable to understand(include) the nature and the purposes of the study, or presenting difficulties of understanding which can compromise the good progress of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
injection Botulinum toxin type-A (BTx-A) | 24 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France